CLINICAL TRIAL: NCT05476458
Title: Prospective, Randomized, Single Center Study to Evaluate Efficacy of Red Dichromatic Imaging (RDI) in Achieving Hemostasis During Peroral Endoscopic Myotomy Using GF 1500 UGI Scope: A Pilot Study
Brief Title: To Evaluate Efficacy of Red Dichromatic Imaging (RDI) in Achieving Hemostasis During POEM Using GF 1500 UGI Scope
Acronym: RDIH-01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Other Study IDs: RDIH-01
Record Dates: First submitted 2022-05-25; First posted 2022-07-27 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: POEMS Syndrome; Hemostatic Disorder
Keywords: Red Dichromatic Imaging; Achieving hemostasis
MeSH Terms: conditions — POEMS Syndrome; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Red Dichromatic Imaging: Per-oral endoscopic myotomy will be performed using novel Evis X1 endoscopy(Olympus corporation, Tokyo, Japan) system. RDI mode 1 and Mode 2 will be used during the procedure. Submucosal bleb will be created by injecting mixture of indigo carmine and normal saline. RDI mode 2 will be used for submucosal injection and Mucosal incision. RDI Mode 2 helps in detection of deep mucosal or submucosal vessels which are the major cause of bleeding. Submucosal dissection and myotomy will be performed under white light. However when there is bleeding, RDI mode 1 will be used for the detection of bleeding point. Bleeding will be controlled with spray coagulation or using Coagrasper. Hemostasis treatment will be performed by switching to RDI only at the time of bleeding during the procedure.
  Interventions: Radiation: Red Light Imaging
- White light imaging: Per-oral endoscopic myotomy will be performed using CV-190 Gastroscope (Olympus corporation, Tokyo, Japan). White light imaging is used during entire procedure. Submucosal bleb will be created by injecting mixture of indigo carmine and normal saline. Initial submucosal injection and Mucosal incision will be performed under white light. RDI Entry point bleed and ease of entry into the tunnel will be marked by trainee at the end of the procedure. Submucosal dissection and myotomy will be performed under white light. When there is bleeding, bleeding point is identified with white light and hemostasis is achieved
  Interventions: Radiation: White Light Imaging

INTERVENTIONS:
Radiation: White Light Imaging — white light imaging is often the preferred option for poem surgery due to its effective results. However, it also comes with some drawbacks that make it difficult to identify areas of bleeding, unlike RDI, WLI cannot enhance the visibility of deep vessels This can lead to longer haemostasis time as the physician must wait for a longer period before stopping the bleeding. This can make it challenging as it may lead to excessive bleeding. This makes RDI a potential solution for those seeking a more accurate approach to treatment.
  Groups: White light imaging
Radiation: Red Light Imaging — Red dichromatic imaging (RDI) is a next-generation image enhancement technique which works by employing green, amber and red wavelengths. Greenlight(520-550nm) can visualize small blood vessels in superficial tissue without extending deep into the mucosa. Amber(595-610nm) and red light (620-640nm) can penetrate deep into the tissue owing to low scattering property. The blood vessels in the deeper tissues absorb the amber light because of strong affinity with hemoglobin. Even though red light can penetrate deep into the tissue, it is weakly absorbed by hemoglobin. Hence the reflected light contains red light and amber light without attenuation.
  Groups: Red Dichromatic Imaging

SUMMARY:
Peroral endoscopic myotomy (POEM) is a novel endoscopic technique for the treatment of achalasia and other esophageal motility disorders. Initially, it was introduced to the world by Inoue et al. in 2008.7 Thereafter; it was rapidly disseminated because of low invasiveness, higher efficacy and technical novelty. The steps of performing POEM include mucosal incision, submucosal tunnel creation, myotomy and closure of the incision. Mucosotomy (2.8%) is the most common adverse event in patients undergoing POEM.8 It can be due to excessive use of cautery because bleeding points could not be seen clearly with white light during active ooze. RDI will help in early recognition of the bleeding points, thus prompt hemostasis. Bleeding during POEM is not very uncommon(0.5-0.7%).9 Early recognition of bleeding points and quicker hemosasis help in decreasing complications. The utility of RDI in the peroral endoscopic myotomy is not studied so far to our knowledge. Hence in this study we would like to look into the utility of red dichromatic imaging in per-oral endoscopic myotomy.

DETAILED DESCRIPTION:
After obtaining departmental and ethics committee clearance, study will be conducted in AIG Hospitals, Hyderabad. Written informed consent will be taken from the patient or relative before enrolling into the study. After enrolment, participants were allocated into Red dichromatic imaging group(Group 1) and White light imaging group(Group 2). All patients will undergo endoscopy prior to the procedure.

All the procedures in this study will be performed by single endoscopic trainee, previously performed less than ten procedures.

Red Dichromatic Imaging (RDI) works by employing green, amber and red wavelength.

* Green light (520-550nm)
* Amber (595-610nm)
* Red Light (620-640nm)

Group 1: Per-oral endoscopic myotomy will be performed using novel Evis X1 endoscopy(Olympus corporation, Tokyo, Japan) system. RDI mode 1 and Mode 2 will be used during the procedure. Submucosal bleb will be created by injecting mixture of indigo carmine and normal saline. RDI mode 2 will be used for submucosal injection and Mucosal incision. RDI Mode 2 helps in detection of deep mucosal or submucosal vessels which are the major cause of bleeding. Submucosal dissection and myotomy will be performed under white light. However when there is bleeding, RDI mode 1 will be used for the detection of bleeding point. Bleeding will be controlled with spray coagulation or using Coagrasper. Hemostasis treatment will be performed by switching to RDI only at the time of bleeding during the procedure.

Group 2: Per-oral endoscopic myotomy will be performed using CV-190 Gastroscope (Olympus corporation, Tokyo, Japan). White light imaging is used during entire procedure. Submucosal bleb will be created by injecting mixture of indigo carmine and normal saline. Initial submucosal injection and Mucosal incision will be performed under white light. RDI Entry point bleed and ease of entry into the tunnel will be marked by trainee at the end of the procedure. Submucosal dissection and myotomy will be performed under white light. When there is bleeding, bleeding point is identified with white light and hemostasis is achieved.

ELIGIBILITY:
Inclusion Criteria:

* • Consecutive consenting patients of both gender posted for POEM in the department of Medical Gastroenterology, AIG Hospitals.

Exclusion Criteria:

* • Patients aged under 18 years of age

  * Unable to provide informed consent
  * Inherited or acquired coagulopathy likely to affect the risk of bleeding
  * Receiving anticoagulant therapy that could not be stopped or bridged prior to procedure
  * Breast feeding, pregnant and lactating women's

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Upto 80 - 100 subjects
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
To determine the change in total procedural time using Red dichromatic imaging (RDI) compared to white light imaging in achieving haemostasis during POEM | To determine the change in total procedural time using Red dichromatic imaging (RDI) compared to white light imaging in achieving haemostasis during POEM
  To determine the change in total procedural time using Red dichromatic imaging (RDI) compared to white light imaging in achieving haemostasis during POEM

SECONDARY OUTCOMES:
To identify avascular mucosal site by identifying and avoiding deep blood vessels using RDI after 1 month and 6 month | Use of RDI in comparison with white light imaging in achieving haemostasis (haemostasis time) after 1 month and 6 months
  Psychological stress experienced by endoscopists during haemostasis treatment as assessed on a scale of 1-5 (1) no stress. (2) minor stress (3) moderate stress (4) high stress (5) very high stress, Ease of mucosal entry by using RDI when compared to white light imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Ramchandani, MBBS, Principal Investigator — Principal Investigator
Locations (2):
- India (2):
  - Aig Hospitals, Hyderabad, Telangana
  - Asian Institute of Gastroenterology, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No